CLINICAL TRIAL: NCT00043420
Title: A Phase I/II Open Label, Multi-Center Study For The Evaluation Of Pf-3512676 (CPG 7909) In Patients With Stage Ib To Iva Cutaneous T-Cell Lymphoma
Brief Title: CPG 7909 in Patients With Cutaneous T-Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C014; CO14, A8501014; NCT00091208 (obsolete NCT alias)
Record Dates: First submitted 2002-08-08; First posted 2002-08-12 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Lymphoma, T-Cell, Cutaneous
Keywords: immunotherapy, lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Lymphoma | interventions — ProMune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Phase I: 0.08 mg/kg (Experimental): Escalating dose groups: 0.08 mg/kg PF-3512676 Injection
  Interventions: Drug: PF-3512676
- Phase I: 0.16 mg/kg (Experimental): Escalating dose groups: 0.16 mg/kg PF-3512676 Injection
  Interventions: Drug: PF-3512676
- Phase I: 0.24 mg/kg (Experimental): Escalating dose groups: 0.24 mg/kg PF-3512676 Injection
  Interventions: Drug: PF-3512676
- Phase I: 0.28 mg/kg (Experimental): Escalating dose groups: 0.28 mg/kg PF-3512676 Injection
  Interventions: Drug: PF-3512676
- Phase I: 0.32 mg/kg (Experimental): Escalating dose groups: 0.32 mg/kg PF-3512676 Injection
  Interventions: Drug: PF-3512676
- Phase I: 0.36 mg/kg (Experimental): Escalating dose groups: 0.36 mg/kg PF-3512676 Injection
  Interventions: Drug: PF-3512676
- Phase II: 10 mg (Experimental): Phase II: 10 mg flat dose (random assignment in Phase II)
  Interventions: Drug: PF-3512676
- Phase II: 25 mg (Experimental): Weekly subcutaneous injections of 25 mg PF-3512676. Treatment continues for a minimum of 8 weeks unless disease progression or unacceptable toxicity occurs, or a maximum of 24 weeks.
  Interventions: Drug: PF-3512676

INTERVENTIONS:
Drug: PF-3512676 — Weekly subcutaneous injections of 0.08mg/kg PF-3512676. Treatment continues for a minimum of 8 weeks unless disease progression or unacceptable toxicity occurs, or a maximum of 24 weeks.
  Other Names: ProMune, CPG 7909
  Arms: Phase I: 0.08 mg/kg
Drug: PF-3512676 — Weekly subcutaneous injections of 0.16mg/kg PF-3512676. Treatment continues for a minimum of 8 weeks unless disease progression or unacceptable toxicity occurs, or a maximum of 24 weeks.
  Other Names: ProMune, CPG 7909
  Arms: Phase I: 0.16 mg/kg
Drug: PF-3512676 — Weekly subcutaneous injections of 0.24mg/kg PF-3512676. Treatment continues for a minimum of 8 weeks unless disease progression or unacceptable toxicity occurs, or a maximum of 24 weeks.
  Other Names: ProMune, CPG 7909
  Arms: Phase I: 0.24 mg/kg
Drug: PF-3512676 — Weekly subcutaneous injections of 0.28mg/kg PF-3512676. Treatment continues for a minimum of 8 weeks unless disease progression or unacceptable toxicity occurs, or a maximum of 24 weeks.
  Other Names: ProMune, CPG 7909
  Arms: Phase I: 0.28 mg/kg
Drug: PF-3512676 — Weekly subcutaneous injections of 0.32mg/kg PF-3512676. Treatment continues for a minimum of 8 weeks unless disease progression or unacceptable toxicity occurs, or a maximum of 24 weeks.
  Other Names: ProMune, CPG 7909
  Arms: Phase I: 0.32 mg/kg
Drug: PF-3512676 — Weekly subcutaneous injections of 0.36mg/kg PF-3512676. Treatment continues for a minimum of 8 weeks unless disease progression or unacceptable toxicity occurs, or a maximum of 24 weeks.
  Other Names: ProMune, CPG 7909
  Arms: Phase I: 0.36 mg/kg
Drug: PF-3512676 — Weekly subcutaneous injections of 10 mg PF-3512676. Treatment continues for a minimum of 8 weeks unless disease progression or unacceptable toxicity occurs, or a maximum of 24 weeks.
  Other Names: ProMune, CPG 7909
  Arms: Phase II: 10 mg
Drug: PF-3512676 — Weekly subcutaneous injections of 25 mg PF-3512676. Treatment continues for a minimum of 8 weeks unless disease progression or unacceptable toxicity occurs, or a maximum of 24 weeks.
  Other Names: ProMune, CPG 7909
  Arms: Phase II: 25 mg

SUMMARY:
To assess the effect of CPG 7909 Injection on Cutaneous T-cell lymphoma and the safety of CPG 7909 Injection in patients with this cancer.

ELIGIBILITY:
Inclusion Criteria:

Patients 18 years or older with biopsy (histopathologically) confirmed cutaneous T-cell lymphoma (limited to mycosis fungoides (MF)) who have had prior therapy with at least one and no more than 3 systemic treatments.

Exclusion Criteria:

Patients with visceral involvement, serious infection or illness including human immunodeficiency virus infection, or a Karnofsky Performance Status (KPS) < 60 will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2003-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Safety: Adverse events, vital signs, clinical and laboratory parameters, physical exams, and ECGs | 24 weeks
Efficacy: Evaluate tumor response as measured by the Composite Assessment of Index Lesion Disease Severity (CA). The primary endpoint will be the overall tumor response rate as assessed by the CA. | 24 weeks

SECONDARY OUTCOMES:
Secondary efficacy endpoints include disease response assessed by the PGA, duration of overall response, duration of CCR, duration of PR, time to response and time to progression of disease. | indeterminate

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- [Derived] Valipour A, Jager M, Wu P, Schmitt J, Bunch C, Weberschock T. Interventions for mycosis fungoides. Cochrane Database Syst Rev. 2020 Jul 7;7(7):CD008946. doi: 10.1002/14651858.CD008946.pub3. PMID 32632956
- [Derived] Kim YH, Girardi M, Duvic M, Kuzel T, Link BK, Pinter-Brown L, Rook AH. Phase I trial of a Toll-like receptor 9 agonist, PF-3512676 (CPG 7909), in patients with treatment-refractory, cutaneous T-cell lymphoma. J Am Acad Dermatol. 2010 Dec;63(6):975-83. doi: 10.1016/j.jaad.2009.12.052. PMID 20888065
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=CO14&StudyName=CPG%207909%20in%20Patients%20With%20Cutaneous%20T-Cell%20Lymphoma